CLINICAL TRIAL: NCT01465659
Title: A Phase I/II Study of the Combination of Temozolomide and Pazopanib in Advanced Pancreatic Neuroendocrine Tumors (PNET)
Brief Title: Temozolomide and Pazopanib Hydrochloride in Treating Patients With Advanced Pancreatic Neuroendocrine Tumors That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other); National Comprehensive Cancer Network (Network); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 11I03; NCI-2011-02939 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00053541 (Other: Northwestern University IRB)
Record Dates: First submitted 2011-10-04; First posted 2011-11-07 (Estimated); Results first posted 2020-06-17 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Pancreatic Alpha Cell Carcinoma; Pancreatic Beta Islet Cell Carcinoma; Pancreatic Delta Cell Carcinoma; Pancreatic G-cell Carcinoma; Recurrent Islet Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Islet Cell | interventions — Temozolomide; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Temozolomide 100 mg/m2 and Pazopanib 400 mg (Experimental): Temozolomide 100 mg/m2 on days 1-7 and 15-21 , Pazopanib 400 mg on days 1-28
  Interventions: Drug: temozolomide; Drug: pazopanib hydrochloride
- Temozolomide 75 mg/m2 and Pazopanib 400 mg (Experimental): Temozolomide 75 mg/m2 on days 1-7 and 15-21 , Pazopanib 400 mg on days 1-28
  Interventions: Drug: temozolomide; Drug: pazopanib hydrochloride
- Temozolomide 150 mg/m2 and Pazopanib 400 mg (Experimental): Temozolomide 150 mg/m2 on days 1-7 and 15-21 , Pazopanib 400 mg on days 1-28
  Interventions: Drug: temozolomide; Drug: pazopanib hydrochloride

INTERVENTIONS:
Drug: temozolomide — Given PO
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Drug: pazopanib hydrochloride — Given PO
  Other Names: GW786034; Votrient

SUMMARY:
This phase I/II trial studies the side effects and best dose of temozolomide and pazopanib hydrochloride when given together and to see how well they work in treating patients with advanced pancreatic neuroendocrine tumors (PNET) that cannot be removed by surgery. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for tumor growth. Giving temozolomide together with pazopanib hydrochloride may be an effective treatment for patients with PNET.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of temozolomide and pazopanib (pazopanib hydrochloride) combination in patients with advanced PNET. (Phase I) II. Determine the overall response rate (ORR). (Phase II)

SECONDARY OBJECTIVES:

I. Determine safety and toxicity profile of the combination of temozolomide and pazopanib in this population. (Phase I) II. Describe the pharmacokinetics of temozolomide alone and in combination with pazopanib. (Phase I) III. Observe the ORR. (Phase I) IV. Determine progression-free survival (PFS) and overall survival (OS), disease control rate (DCR), and duration of response (DOR). (Phase II) V. Determine the safety and toxicity profile of the combination in a larger cohort of patients. (Phase II)

TERTIARY OBJECTIVES:

I. Examine the relationship between tumor blood flow, as measured by perfusion functional computed tomography (f CT), and overall response.

II. Correlate the expression of tissue methyl-guanine methyl transferase (MGMT) as measured by immunohistochemistry (IHC) with ORR and PFS.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive temozolomide orally (PO) once daily (QD) on days 1-7 and 15-21 and pazopanib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed islet cell carcinoma (PNET) not amenable to surgical resection
* Patients may have had 0-2 prior therapies; prior chemoembolization or local ablative therapies are permitted if completed >= 6 weeks prior to study enrollment
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must have a life expectancy > 3 months
* Patients must have radiographically measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria
* Patients' baseline blood pressure must be adequately controlled with or without antihypertensive medications prior to enrollment (systolic < 140 mmHg, diastolic < 90 mmHg)
* Patients must have left ventricular ejection fraction (LVEF) >= 50 as measured by echocardiogram or multi gated acquisition scan (MUGA)
* Absolute neutrophil count (ANC) >= 1,500/µL
* Platelets >= 100,000/µL
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 2 mg/dL or =< 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 5 times ULN
* International normalized ratio (INR) =< 1.2 times upper limit of normal (ULN); subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation
* Activated partial thromboplastin time (aPTT) =< 1.2 x ULN
* Albumin >= 2.8 g/dL
* Serum creatinine =< 1.5 times ULN OR if serum creatinine >= 1.5 mg/dL, calculated creatinine clearance >= 30 mL/min
* Urine protein to creatinine ratio < 1 OR 24-hour urine protein < 1 g
* Patients must be able to tolerate oral medications
* Females of child-bearing potential must have a negative pregnancy test within 14 days of study enrollment and must agree to use an effective method of birth control during treatment and for three months after receiving their last dose of study drug; males must agree to use an effective method of birth control during treatment and for three months after receiving their last dose of study drug; all patients must notify treating provider immediately if any suspicion of pregnancy or conception;
* Child-bearing potential is defined as any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: has NOT undergone a hysterectomy or bilateral oophorectomy; OR has NOT been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* The eligibility of patients receiving any medications or substances known or with potential to affect the activity or pharmacokinetics of temozolomide and/or pazopanib will be determined following review of the case by the Principal Investigator and the Data Monitoring Committee (DMC); efforts should be made to switch patients who are taking enzyme-inducing agents to other medications
* Patients must have given signed, informed consent prior to registration on study

Exclusion Criteria:

* Patients taking immunosuppressive medications (including systemic corticosteroids unless used for adrenal replacement), appetite stimulants, acute therapy for asthma or acute bronchitis exacerbation, or antiemetics are NOT eligible for participation
* Patients with known human immunodeficiency virus (HIV) infection are NOT eligible for participation
* Patients with uncontrolled hypertension (>= 140/90 mmHg) are NOT eligible for participation
* Patients with uncontrolled hyperlipidemia (total cholesterol > 350 or triglycerides > 300) are NOT eligible for participation
* Patients who have had a transfusion within 7 days of screening are NOT eligible for participation
* Patients with symptomatic brain or bone metastasis (mets) are NOT eligible for participation; prior radiation and/or steroid therapy for brain or bone mets must be completed >= 2 weeks prior to study enrollment
* Patients with a history of seizure disorder requiring antiepileptic medication or brain metastases with seizures are NOT eligible for participation
* Patients with an active second malignancy (other than non-melanoma skin cancer or cervical carcinoma in situ) are NOT eligible for participation; patients who have a history of malignancy are not considered to have a currently active malignancy if they have completed therapy and are now considered by their physician to be at < 30% risk for relapse
* Patients with clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding are NOT eligible for participation; these may include (but are not limited to):
* Active peptic ulcer disease
* Known intraluminal metastatic lesion/s with risk of bleeding
* Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease)
* Other gastrointestinal conditions with increased risk of perforation
* Patients with a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment are NOT eligible for participation
* Patients with clinically significant gastrointestinal abnormalities that may affect absorption of the investigational product including are NOT eligible for participation; these may include (but are not limited to):
* Malabsorption syndrome
* Major resection of the stomach or small bowel
* Patients with a history of any one or more of the following cardiovascular conditions within the past 6 months prior to study enrollment are NOT eligible for participation:
* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* Coronary artery bypass graft surgery
* Symptomatic peripheral vascular disease
* Class III or IV congestive heart failure, as defined by the New York Heart Association
* Patients with a corrected QT interval (QTc) > 480 msecs are NOT eligible for participation
* Patients with a history of transient ischemic attack (TIA) or cerebrovascular accident (CVA) within the past 6 months prior to study enrollment are NOT eligible for participation
* Patients with a history of any one or more of the following thromboembolic events within the past 6 months prior to study enrollment are NOT eligible for participation:
* Pulmonary embolism
* Untreated deep venous thrombosis (DVT); subjects with recent DVT who have been therapeutically coagulated for at least 6 weeks ARE eligible
* Patients who have undergone major surgery or trauma within 28 days prior to the first dose of investigational product and/or present with any non-healing wound, fracture, or ulcer are NOT eligible for participation; procedures such as catheter placement not considered to be major surgery
* Patients with known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage are NOT eligible for participation
* Lesions infiltrating major pulmonary vessels (contiguous tumor and vessels) are excluded; however, the presence of a tumor that is touching, but not infiltrating, the vessels is acceptable; CT with contrast is strongly recommended to evaluate such lesions
* Large protruding endobronchial lesions in the main or lobar bronchi are excluded; however, endobronchial lesions in the segmented bronchi are allowed
* Lesions extensively infiltrating the main or lobar bronchi are excluded; however, minor infiltrations in the wall of the bronchi are allowed
* Patients who have had recent hemoptysis (>= 1/2 teaspoon of red blood within 8 weeks before first dose of study drug) are NOT eligible for participation
* Patients who have any history of allergic reaction(s) attributed to compounds of similar composition to temozolomide, pazopanib, their metabolites, or any component of their formulation are NOT eligible for participation
* Females who are pregnant or lactating, fertile males, or females of child-bearing potential who are not willing to comply with an effective double method of birth control are NOT eligible for participation
* Patients with a psychiatric illness, other condition or significant medical illness, or social situation which, in the investigator's opinion, would limit compliance or ability to comply with study requirements are NOT eligible for participation
* Patients who have taken medications that are known strong inducers or inhibitors of Cytochrome P450 3A4 (CYP3A4) within 28 days prior to registration are NOT eligible for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-12-12 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2021-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Halla Nimeiri, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was opened to enrollment on November 15th 2011 with the first patient starting treatment December 12th 2011. The study was designed to enroll up to 40 patients with a phase I dose escalation portion and a phase II expansion portion at the determined dose. The study was closed to further enrollment February 27 2019.
Groups:
- Cohort 1 - Temozolomide 150 mg/m2 and Pazopanib 400 mg: Temozolomide 150 mg/m2 on days 1-7 and 15-21 , Pazopanib 400 mg on days 1-28
  temozolomide: Given PO
  pazopanib hydrochloride: Given PO
- Cohort -1 -Temozolomide 100 mg/m2 and Pazopanib 400 mg: Temozolomide 100 mg/m2 on days 1-7 and 15-21 , Pazopanib 400 mg on days 1-28
  temozolomide: Given PO
  pazopanib hydrochloride: Given PO
- Cohort -2 - Temozolomide 75 mg/m2 and Pazopanib 400 mg: Temozolomide 75 mg/m2 on days 1-7 and 15-21 , Pazopanib 400 mg on days 1-28
  temozolomide: Given PO
  pazopanib hydrochloride: Given PO
- Phase II -Temozolomide 75 mg/m2 and Pazopanib 400 mg: Temozolomide 75mg/m2 on days 1-7 and 15-21 , Pazopanib 400 mg on days 1-28
  temozolomide: Given PO
  pazopanib hydrochloride: Given PO
Period: Completed 1 Cycle of Treatment
Arm/Group | Cohort 1 - Temozolomide 150 mg/m2 and Pazopanib 400 mg | Cohort -1 -Temozolomide 100 mg/m2 and Pazopanib 400 mg | Cohort -2 - Temozolomide 75 mg/m2 and Pazopanib 400 mg | Phase II -Temozolomide 75 mg/m2 and Pazopanib 400 mg
Started | 7 | 5 | 6 | 11
Completed 1 Cycle of Treatment | 7 | 4 | 6 | 11
Completed | 7 | 4 | 6 | 10
Not Completed | 0 | 1 | 0 | 1
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Completed 2 Cycles/Reached 1st Response
Arm/Group | Cohort 1 - Temozolomide 150 mg/m2 and Pazopanib 400 mg | Cohort -1 -Temozolomide 100 mg/m2 and Pazopanib 400 mg | Cohort -2 - Temozolomide 75 mg/m2 and Pazopanib 400 mg | Phase II -Temozolomide 75 mg/m2 and Pazopanib 400 mg
Started | 7 | 4 | 6 | 10
Attempted 2 Cycles of Treatment | 7 | 4 | 6 | 10
Reached 1st Response | 7 | 4 | 6 | 10
Assessed to Move on to Next Cycle | 7 | 4 | 4 | 10
Completed | 5 | 4 | 4 | 9
Not Completed | 2 | 0 | 2 | 1
Not completed — Progressive Disease | 1 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 0
Period: Went on to Cycle 3 and Beyond
Arm/Group | Cohort 1 - Temozolomide 150 mg/m2 and Pazopanib 400 mg | Cohort -1 -Temozolomide 100 mg/m2 and Pazopanib 400 mg | Cohort -2 - Temozolomide 75 mg/m2 and Pazopanib 400 mg | Phase II -Temozolomide 75 mg/m2 and Pazopanib 400 mg
Started | 5 | 4 | 4 | 9
Completed | 5 | 4 | 4 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Completed Follow for 1 Year
Arm/Group | Cohort 1 - Temozolomide 150 mg/m2 and Pazopanib 400 mg | Cohort -1 -Temozolomide 100 mg/m2 and Pazopanib 400 mg | Cohort -2 - Temozolomide 75 mg/m2 and Pazopanib 400 mg | Phase II -Temozolomide 75 mg/m2 and Pazopanib 400 mg
Started (Any patient that is treated with study drug goes into follow up after treatment discontinuation.) | 7 | 4 | 6 | 11
Completed | 1 | 1 | 4 | 7
Not Completed | 6 | 3 | 2 | 4
Not completed — Death | 6 | 3 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Temozolomide 150 mg/m2 and Pazopanib 400 mg | Cohort -1 -Temozolomide 100 mg/m2 and Pazopanib 400 mg | Cohort -2 - Temozolomide 75 mg/m2 and Pazopanib 400 mg | Phase II -Temozolomide 75 mg/m2 and Pazopanib 400 mg | Total
Number analyzed (Participants) | 7 | 5 | 6 | 11 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 6 | 9 | 25
  >=65 years | 0 | 2 | 0 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 6 | 13
  Male | 4 | 3 | 4 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 6 | 5 | 6 | 9 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 6 | 5 | 6 | 10 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 6 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: Determine the Maximum Tolerated Dose (MTD) of Temozolomide in Combination With 400 mg Pazopanib in Patients With Advanced Pancreatic Neuroendocrine Tumor (PNET) in Phase I
Description: MTD and recommended phase II dose (RP2D) determination for the combination of temozolomide in combination with 400mg pazopanib in patients with advanced PNET will be achieved using a standard "3+3" dose escalation/de-escalation design. After each 3 patients are enrolled into the study, further enrollment will be temporarily suspended until safety has been reviewed for the first 28 days of treatment to determine if dose limiting toxicities have been experienced by patients and if a further 3 patients should be enrolled at the current dose or dose escalation/de-escalation for the next 3 patients should occur.
Time Frame: After 28 days (1 cycle of treatment)
Population: 1 patient in Cohort -1 was not evaluable for this endpoint due to inability to absorb oral medications secondary to bowel edema
Measure: Number; unit: mg/m2
Groups:
- Cohort 1/Cohort -1/Cohort -2 - Temozolomide and Pazopanib: Temozolomide 75 - 150 mg/m2 on days 1-7 and 15-21 , Pazopanib 400 mg on days 1-28
  temozolomide: Given PO
  pazopanib hydrochloride: Given PO
Arm/Group | Cohort 1/Cohort -1/Cohort -2 - Temozolomide and Pazopanib
Number analyzed (Participants) | 17
mg/m2 | 75

2. Primary Outcome: Overall Response Rate (ORR) in Patients With Advanced Neuroendocrine Tumors (PNET) Treated With Temozolomide and Pazopanib Combination Treatment at the RP2D in Phase II
Description: Overall response rate will be determined by the number of patients who's best response as assessed by RECIST 1.1 is complete response (CR) and partial response (PR) in patients with PNET that are enrolled at the recommended phase II dose (RP2D) (PK cohort included).
  CR= Disappearance of all target lesions PR = At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: After two cycles of treatment (8 weeks)
Population: 1 patient was determined not to be evaluable for response in phase II
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II -Temozolomide 75 mg/m2 and Pazopanib 400 mg
Number analyzed (Participants) | 10
Participants | 0

3. Secondary Outcome: Number of Patients Who Experience Toxicity Events Undergoing This Treatment.
Description: Safety and toxicity will be reported in the number of patients who experience adverse events during treatment, graded using CTCAE 4.03.
  In general the severity of an AE is graded as follows:
  Mild (grade 1): the event causes discomfort without disruption of normal daily activities.
  Moderate (grade 2): the event causes discomfort that affects normal daily activities.
  Severe (grade 3): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status.
  Life-threatening (grade 4): the patient was at risk of death at the time of the event. Fatal (grade 5): the event caused death.
Time Frame: During treatment and up to one month post last dose of study drug. Range of cycles completed by patients was 1-41 where one cycle =28 days.
Measure: Number; unit: patients
Arm/Group | Cohort 1 - Temozolomide 150 mg/m2 and Pazopanib 400 mg | Cohort -1 -Temozolomide 100 mg/m2 and Pazopanib 400 mg | Cohort -2 - Temozolomide 75 mg/m2 and Pazopanib 400 mg | Phase II -Temozolomide 75 mg/m2 and Pazopanib 400 mg
Number analyzed (Participants) | 7 | 5 | 6 | 11
patients
  Any AE | 7 | 5 | 6 | 11
  AE related to treatment | 7 | 5 | 6 | 11
  SAE | 3 | 3 | 1 | 1
  SAE related to treatment | 3 | 1 | 1 | 1
  Grade 5 SAE | 0 | 1 | 0 | 0
  Came off treatment due to an AE | 3 | 3 | 3 | 2

4. Secondary Outcome: Plasma Temozolomide Concentration in the Blood at Various Timepoints After Administration
Description: For the Six Patients in Phase I portion who are enrolled in the PK cohort: Blood will be drawn on Day 1 before beginning treatment and again at 10 minutes, 30 minutes, 1, 2, 3, 4, 6 and 8 hours after beginning treatment. On Day 2- 24 hours after the first dose from Day 1, and again 10 minutes, 30 minutes, 1, 2, 3, 4, 6 and 8 hours after taking the second dose. Day 3 - 24 hours after the second dose from Day 2.
  Cycle 1 Day 1 only temozolomide will be taken by the patient and on Cycle 2 Day 2, temozolomide and pazopanib will be taken by the patient. Data that was collected but not analyzed. The data that was collected is reported below in raw form.
Time Frame: Multiple timepoints during Days 1-3 of cycle 1 and cycle 2 (1 cycle =28 days)
Population: Data that was collected but not analyzed. The data that was collected is reported below for each patient at each timepoint.
Measure: Number; unit: ng/mL
Groups:
- Temozolomide 75 mg/m2 and Pazopanib 400 mg: Temozolomide 75mg/m2 on days 1-7 and 15-21 , Pazopanib 400 mg on days 1-28
  temozolomide: Given PO
  pazopanib hydrochloride: Given PO
Arm/Group | Temozolomide 75 mg/m2 and Pazopanib 400 mg
Number analyzed (Participants) | 6
ng/mL
  Patient #1 : Cycle 1 Day 1 at time 0 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 1 Day 1 at time 0 hours | 0
  Patient #1 : Cycle 1 Day 1 at time 0.17 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 1 Day 1 at time 0.17 hours | 0
  Patient #1 : Cycle 1 Day 1 at time 0.5 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 1 Day 1 at time 0.5 hours | 91.8
  Patient #1 : Cycle 1 Day 1 at time 1 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 1 Day 1 at time 1 hours | 425.5
  Patient #1 : Cycle 1 Day 1 at time 2 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 1 Day 1 at time 2 hours | 462
  Patient #1 : Cycle 1 Day 1 at time 3 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 1 Day 1 at time 3 hours | 583
  Patient #1 : Cycle 1 Day 1 at time 4 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 1 Day 1 at time 4 hours | 210.5
  Patient #1 : Cycle 1 Day 1 at time 6 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 1 Day 1 at time 6 hours | 105
  Patient #1 : Cycle 1 Day 1 at time 8 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 1 Day 1 at time 8 hours | 44
  Patient #1 : Cycle 1 Day 1 at time 24 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 1 Day 1 at time 24 hours | 0
  Patient #1 : Cycle 2 Day 1 at time 0 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 2 Day 1 at time 0 hours | 0
  Patient #1 : Cycle 2 Day 1 at time 0.17 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 2 Day 1 at time 0.17 hours | 0
  Patient #1 : Cycle 2 Day 1 at time 0.5 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 2 Day 1 at time 0.5 hours | 25.2
  Patient #1 : Cycle 2 Day 1 at time 1 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 2 Day 1 at time 1 hours | 90.8
  Patient #1 : Cycle 2 Day 1 at time 2 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 2 Day 1 at time 2 hours | 516.5
  Patient #1 : Cycle 2 Day 1 at time 3 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 2 Day 1 at time 3 hours | 255
  Patient #1 : Cycle 2 Day 1 at time 4 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 2 Day 1 at time 4 hours | 519
  Patient #1 : Cycle 2 Day 1 at time 6 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 2 Day 1 at time 6 hours | 154
  Patient #1 : Cycle 2 Day 1 at time 8 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 2 Day 1 at time 8 hours | 99.9
  Patient #1 : Cycle 2 Day 1 at time 24 hours: number analyzed (Participants) | 1
  Patient #1 : Cycle 2 Day 1 at time 24 hours | 0
  Patient #2 : Cycle 1 Day 1 at time 0 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 1 Day 1 at time 0 hours | 0
  Patient #2 : Cycle 1 Day 1 at time 0.17 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 1 Day 1 at time 0.17 hours | 0
  Patient #2 : Cycle 1 Day 1 at time 0.5 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 1 Day 1 at time 0.5 hours | 54.9
  Patient #2 : Cycle 1 Day 1 at time 1 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 1 Day 1 at time 1 hours | 494
  Patient #2 : Cycle 1 Day 1 at time 2 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 1 Day 1 at time 2 hours | 660.5
  Patient #2 : Cycle 1 Day 1 at time 3 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 1 Day 1 at time 3 hours | 557.5
  Patient #2 : Cycle 1 Day 1 at time 4 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 1 Day 1 at time 4 hours | 99
  Patient #2 : Cycle 1 Day 1 at time 6 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 1 Day 1 at time 6 hours | 105.5
  Patient #2 : Cycle 1 Day 1 at time 8 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 1 Day 1 at time 8 hours | 109.5
  Patient #2 : Cycle 1 Day 1 at time 24 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 1 Day 1 at time 24 hours | 0
  Patient #2 : Cycle 2 Day 1 at time 0 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 2 Day 1 at time 0 hours | 0
  Patient #2 : Cycle 2 Day 1 at time 0.17 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 2 Day 1 at time 0.17 hours | 0
  Patient #2 : Cycle 2 Day 1 at time 0.5 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 2 Day 1 at time 0.5 hours | 41.6
  Patient #2 : Cycle 2 Day 1 at time 1 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 2 Day 1 at time 1 hours | 115
  Patient #2 : Cycle 2 Day 1 at time 2 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 2 Day 1 at time 2 hours | 1490
  Patient #2 : Cycle 2 Day 1 at time 3 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 2 Day 1 at time 3 hours | 961.5
  Patient #2 : Cycle 2 Day 1 at time 4 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 2 Day 1 at time 4 hours | 382.5
  Patient #2 : Cycle 2 Day 1 at time 6 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 2 Day 1 at time 6 hours | 510.5
  Patient #2 : Cycle 2 Day 1 at time 8 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 2 Day 1 at time 8 hours | 109.5
  Patient #2 : Cycle 2 Day 1 at time 24 hours: number analyzed (Participants) | 1
  Patient #2 : Cycle 2 Day 1 at time 24 hours | 0
  Patient #3 : Cycle 1 Day 1 at time 0 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 1 Day 1 at time 0 hours | 0
  Patient #3 : Cycle 1 Day 1 at time 0.17 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 1 Day 1 at time 0.17 hours | 0
  Patient #3 : Cycle 1 Day 1 at time 0.5 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 1 Day 1 at time 0.5 hours | 527
  Patient #3 : Cycle 1 Day 1 at time 1 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 1 Day 1 at time 1 hours | 1670
  Patient #3 : Cycle 1 Day 1 at time 2 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 1 Day 1 at time 2 hours | 2440
  Patient #3 : Cycle 1 Day 1 at time 3 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 1 Day 1 at time 3 hours | 2024
  Patient #3 : Cycle 1 Day 1 at time 4 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 1 Day 1 at time 4 hours | 1466
  Patient #3 : Cycle 1 Day 1 at time 6 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 1 Day 1 at time 6 hours | 718
  Patient #3 : Cycle 1 Day 1 at time 8 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 1 Day 1 at time 8 hours | 317
  Patient #3 : Cycle 1 Day 1 at time 24 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 1 Day 1 at time 24 hours | 4.3
  Patient #3 : Cycle 2 Day 1 at time 0 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 2 Day 1 at time 0 hours | 4.1
  Patient #3 : Cycle 2 Day 1 at time 0.17 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 2 Day 1 at time 0.17 hours | 241
  Patient #3 : Cycle 2 Day 1 at time 0.5 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 2 Day 1 at time 0.5 hours | 909
  Patient #3 : Cycle 2 Day 1 at time 1 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 2 Day 1 at time 1 hours | 2130
  Patient #3 : Cycle 2 Day 1 at time 2 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 2 Day 1 at time 2 hours | 2490
  Patient #3 : Cycle 2 Day 1 at time 3 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 2 Day 1 at time 3 hours | 1933
  Patient #3 : Cycle 2 Day 1 at time 4 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 2 Day 1 at time 4 hours | 1586
  Patient #3 : Cycle 2 Day 1 at time 6 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 2 Day 1 at time 6 hours | 761
  Patient #3 : Cycle 2 Day 1 at time 8 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 2 Day 1 at time 8 hours | 328
  Patient #3 : Cycle 2 Day 1 at time 24 hours: number analyzed (Participants) | 1
  Patient #3 : Cycle 2 Day 1 at time 24 hours | 4.75
  Patient #4 : Cycle 1 Day 1 at time 0 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 1 Day 1 at time 0 hours | 0
  Patient #4 : Cycle 1 Day 1 at time 0.17 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 1 Day 1 at time 0.17 hours | 3.6
  Patient #4 : Cycle 1 Day 1 at time 0.5 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 1 Day 1 at time 0.5 hours | 492
  Patient #4 : Cycle 1 Day 1 at time 1 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 1 Day 1 at time 1 hours | 3025
  Patient #4 : Cycle 1 Day 1 at time 2 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 1 Day 1 at time 2 hours | 2805
  Patient #4 : Cycle 1 Day 1 at time 3 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 1 Day 1 at time 3 hours | 1765
  Patient #4 : Cycle 1 Day 1 at time 4 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 1 Day 1 at time 4 hours | 1430
  Patient #4 : Cycle 1 Day 1 at time 6 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 1 Day 1 at time 6 hours | 686.5
  Patient #4 : Cycle 1 Day 1 at time 8 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 1 Day 1 at time 8 hours | 383
  Patient #4 : Cycle 1 Day 1 at time 24 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 1 Day 1 at time 24 hours | 1.2
  Patient #4 : Cycle 2 Day 1 at time 0 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 2 Day 1 at time 0 hours | 2.4
  Patient #4 : Cycle 2 Day 1 at time 0.17 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 2 Day 1 at time 0.17 hours | 2.3
  Patient #4 : Cycle 2 Day 1 at time 0.5 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 2 Day 1 at time 0.5 hours | 3.0
  Patient #4 : Cycle 2 Day 1 at time 1 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 2 Day 1 at time 1 hours | 1.6
  Patient #4 : Cycle 2 Day 1 at time 2 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 2 Day 1 at time 2 hours | 1.0
  Patient #4 : Cycle 2 Day 1 at time 3 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 2 Day 1 at time 3 hours | 12
  Patient #4 : Cycle 2 Day 1 at time 4 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 2 Day 1 at time 4 hours | 3360
  Patient #4 : Cycle 2 Day 1 at time 6 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 2 Day 1 at time 6 hours | 2610
  Patient #4 : Cycle 2 Day 1 at time 8 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 2 Day 1 at time 8 hours | 1225
  Patient #4 : Cycle 2 Day 1 at time 24 hours: number analyzed (Participants) | 1
  Patient #4 : Cycle 2 Day 1 at time 24 hours | 3285
  Patient #5 : Cycle 1 Day 1 at time 0 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 1 Day 1 at time 0 hours | 0
  Patient #5 : Cycle 1 Day 1 at time 0.17 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 1 Day 1 at time 0.17 hours | 19.1
  Patient #5 : Cycle 1 Day 1 at time 0.5 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 1 Day 1 at time 0.5 hours | 177
  Patient #5 : Cycle 1 Day 1 at time 1 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 1 Day 1 at time 1 hours | 227
  Patient #5 : Cycle 1 Day 1 at time 2 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 1 Day 1 at time 2 hours | 275
  Patient #5 : Cycle 1 Day 1 at time 3 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 1 Day 1 at time 3 hours | 829.5
  Patient #5 : Cycle 1 Day 1 at time 4 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 1 Day 1 at time 4 hours | 925
  Patient #5 : Cycle 1 Day 1 at time 6 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 1 Day 1 at time 6 hours | 1145
  Patient #5 : Cycle 1 Day 1 at time 8 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 1 Day 1 at time 8 hours | 819.5
  Patient #5 : Cycle 1 Day 1 at time 24 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 1 Day 1 at time 24 hours | 44.2
  Patient #5 : Cycle 2 Day 1 at time 0 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 2 Day 1 at time 0 hours | 0
  Patient #5 : Cycle 2 Day 1 at time 0.17 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 2 Day 1 at time 0.17 hours | 108
  Patient #5 : Cycle 2 Day 1 at time 0.5 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 2 Day 1 at time 0.5 hours | 166.5
  Patient #5 : Cycle 2 Day 1 at time 1 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 2 Day 1 at time 1 hours | 188.5
  Patient #5 : Cycle 2 Day 1 at time 2 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 2 Day 1 at time 2 hours | 422.5
  Patient #5 : Cycle 2 Day 1 at time 3 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 2 Day 1 at time 3 hours | 716.5
  Patient #5 : Cycle 2 Day 1 at time 4 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 2 Day 1 at time 4 hours | 1070
  Patient #5 : Cycle 2 Day 1 at time 6 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 2 Day 1 at time 6 hours | 1180
  Patient #5 : Cycle 2 Day 1 at time 8 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 2 Day 1 at time 8 hours | 744.5
  Patient #5 : Cycle 2 Day 1 at time 24 hours: number analyzed (Participants) | 1
  Patient #5 : Cycle 2 Day 1 at time 24 hours | 36.7
  Patient #6a : Cycle 1 Day 1 at time 0 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 1 Day 1 at time 0 hours | 0
  Patient #6a : Cycle 1 Day 1 at time 0.17 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 1 Day 1 at time 0.17 hours | 459.5
  Patient #6a : Cycle 1 Day 1 at time 0.5 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 1 Day 1 at time 0.5 hours | 3055
  Patient #6a : Cycle 1 Day 1 at time 1 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 1 Day 1 at time 1 hours | 2720
  Patient #6a : Cycle 1 Day 1 at time 2 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 1 Day 1 at time 2 hours | 1735
  Patient #6a : Cycle 1 Day 1 at time 3 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 1 Day 1 at time 3 hours | 1470
  Patient #6a : Cycle 1 Day 1 at time 4 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 1 Day 1 at time 4 hours | 1195
  Patient #6a : Cycle 1 Day 1 at time 6 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 1 Day 1 at time 6 hours | 499.5
  Patient #6a : Cycle 1 Day 1 at time 8 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 1 Day 1 at time 8 hours | 251
  Patient #6a : Cycle 1 Day 1 at time 24 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 1 Day 1 at time 24 hours | 1.5
  Patient #6a : Cycle 2 Day 1 at time 0 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 2 Day 1 at time 0 hours | 0
  Patient #6a : Cycle 2 Day 1 at time 0.17 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 2 Day 1 at time 0.17 hours | 67.7
  Patient #6a : Cycle 2 Day 1 at time 0.5 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 2 Day 1 at time 0.5 hours | 4095
  Patient #6a : Cycle 2 Day 1 at time 1 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 2 Day 1 at time 1 hours | 2135
  Patient #6a : Cycle 2 Day 1 at time 2 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 2 Day 1 at time 2 hours | 2095
  Patient #6a : Cycle 2 Day 1 at time 3 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 2 Day 1 at time 3 hours | 1445
  Patient #6a : Cycle 2 Day 1 at time 4 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 2 Day 1 at time 4 hours | 1025.5
  Patient #6a : Cycle 2 Day 1 at time 6 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 2 Day 1 at time 6 hours | 324.5
  Patient #6a : Cycle 2 Day 1 at time 8 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 2 Day 1 at time 8 hours | 192.5
  Patient #6a : Cycle 2 Day 1 at time 24 hours: number analyzed (Participants) | 1
  Patient #6a : Cycle 2 Day 1 at time 24 hours | 1.3

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS will be defined as will be defined as the time from the first study treatment to the first occurrence of progression or death. Progressive disease will be assessed using RECIST v1.1 criteria where in general the following definition is true: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum recorded on study AND an absolute increase in the sum of at least 5 mm OR the appearance of one or more new lesions
Time Frame: Baseline and after every 2 cycles of treatment (8 weeks) for up to 40 months
Population: The study did not reach its anticipated sample size and anticipated endpoints for phase II. Due to this and relatively small number of patients it was determined by the PI to have no merit or statistical significance to calculate PFS per dose cohort and dose cohorts were combined to summarize PFS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1/Cohort -1/Cohort -2 - Temozolomide and Pazopanib
Number analyzed (Participants) | 29
months | 9.38 [6.18 to 13.3]

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first study treatment until death from any cause.
Time Frame: Baseline and after every 2 cycles of treatment (8 weeks) and up to 60 months
Population: The study did not reach its anticipated sample size and anticipated endpoints for phase II. Due to this and relatively small number of patients it was determined by the PI to have no merit or statistical significance to calculate OS per dose cohort and dose cohorts were combined to summarize OS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1/Cohort -1/Cohort -2 - Temozolomide and Pazopanib
Number analyzed (Participants) | 29
months | 24.2 [18.3 to NA] — Upper limit was not reached

7. Secondary Outcome: Number of Patients Experiencing Response to Treatment or Stable Disease (Disease Control Rate)
Description: Disease Control Rate (DCR) is defined as the number of patients demonstrating the complete response, partial response or stable disease.
  In general the following is true:
  Complete Response (CR) Disappearance of all target lesions. Disappearance of all non-target lesions and normalization of tumor marker level.
  Partial Response (PR) At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters Stable Disease (SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of diameters while on study
Time Frame: After every 2 courses of treatment (8 weeks) for up to 41 cycles where 1 cycle =28 days.
Population: The study did not reach its anticipated sample size and anticipated endpoints for phase II. Due to this and relatively small number of patients it was determined by the PI to have no merit or statistical significance to calculate DCR per dose cohort and dose cohorts were combined to summarize DCR.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1/Cohort -1/Cohort -2 - Temozolomide and Pazopanib
Number analyzed (Participants) | 29
Participants | 20

8. Secondary Outcome: Number of Months That Patients Maintain a Response to Treatment Until Disease Progression or Death (Duration of Response)
Description: Duration of response (DOR) is defined at the time from documented overall response (compete response, partial response, stable disease) until disease progression where the following are true:
  Complete Response (CR) Disappearance of all target lesions. Disappearance of all non-target lesions and normalization of tumor marker level.
  Partial Response (PR) At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters Stable Disease (SD) Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of diameters while on study
Time Frame: After every 2 courses of treatment (8 weeks)
Population: Data not collected or analyzed for this outcome measure
Arm/Group | Cohort 1/Cohort -1/Cohort -2 - Temozolomide and Pazopanib
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Determine the Relationship Between Tumor Blood Flow and Overall Response Rate
Description: For Patients in Phase II Portion: Patients will have a perfusion functional computed tomography (fCT) scan at baseline and after two courses of treatment.
Time Frame: At Baseline and after two corurses of treatment (8 weeks)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Amount of a Particular Tumor Biomarker in Blood as Correlated With Progression Free Survival
Description: For Patients in Phase II Portion: The level of expression of tissue methyl-guanine methytransferase (MGMT)will be measured in tissue from the diagnostic biopsy and these results will be correlated with response rate.
Time Frame: Baseline and at Response assessment after two courses of treatment (8 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Patients were monitored for adverse events for the duration of treatment and up to 1 month post last dose of study drug. Range of cycles completed by patients was 1-41 where one cycle =28 days
Description: This contains data that has been collected and reported in the eCRFs on April 22nd 2020 and may be updated at the time of secondary outcome measure reporting. Due to the way that adverse events and serious adverse events are collect and reported in the eCRFs the "other" adverse events may contain some serious adverse event data.
Arm/Group | Cohort 1 - Temozolomide 150 mg/m2 and Pazopanib 400 mg | Cohort -1 -Temozolomide 100 mg/m2 and Pazopanib 400 mg | Cohort -2 - Temozolomide 75 mg/m2 and Pazopanib 400 mg | Phase II -Temozolomide 75 mg/m2 and Pazopanib 400 mg
All-Cause Mortality (participants affected / at risk) | 6/7 | 4/5 | 2/6 | 4/11
Serious Adverse Events (participants affected / at risk) | 3/7 | 3/5 | 1/6 | 1/11
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5 | 6/6 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Temozolomide 150 mg/m2 and Pazopanib 400 mg (N=7) | Cohort -1 -Temozolomide 100 mg/m2 and Pazopanib 400 mg (N=5) | Cohort -2 - Temozolomide 75 mg/m2 and Pazopanib 400 mg (N=6) | Phase II -Temozolomide 75 mg/m2 and Pazopanib 400 mg (N=11)
Upper Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Shingles (Infections and infestations) | 1 (1) | 0 | 0 | 0
Guillian-Barre Syndrome (General disorders) | 1 (1) | 0 | 0 | 0
ACTH secreting tumor with cushings syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (2) | 0 | 0 — patient with hypokalemia and diarrhea during first event and thrombocytopenia and leukopenia during the second event
AST and ALT increased (Investigations) | 0 | 1 (1) | 1 (1) | 0
Thrombocytopenia (Investigations) | 1 (1) | 0 | 0 | 0 — Patient also with neutropenia and white blood cell decreased during this event
Epistasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 0
Splenic hemorrage (Blood and lymphatic system disorders) | 1 (1) | 0 | 0 | 0
Protein calorie malnutrition (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 0 — Patient also with diarrhea at the time
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Temozolomide 150 mg/m2 and Pazopanib 400 mg (N=7) | Cohort -1 -Temozolomide 100 mg/m2 and Pazopanib 400 mg (N=5) | Cohort -2 - Temozolomide 75 mg/m2 and Pazopanib 400 mg (N=6) | Phase II -Temozolomide 75 mg/m2 and Pazopanib 400 mg (N=17)
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Hemoglobin (anemia) (Blood and lymphatic system disorders) | 6 | 4 | 3 | 6
Petechiae (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Red blood cells decreased (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Increased heart rate (Cardiac disorders) | 1 | 0 | 0 | 0
Chest pain (Cardiac disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 1
Edema limbs (General disorders) | 1 | 1 | 3 | 3
Fatigue (General disorders) | 5 | 3 | 4 | 4
Fever (General disorders) | 1 | 0 | 0 | 1
Injection site reaction (General disorders) | 1 | 0 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 3 | 0 | 0 | 1
Pain (General disorders) | 3 | 0 | 1 | 1
Night sweats (General disorders) | 1 | 0 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 1 | 0
Localized edema (General disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Poison ivy rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hair color changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Precancerous lesion on lip/face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin discoloration post shingles (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Petechial rash on breasts (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ulceration on lower lip (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hair color lightening (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Excoriations anterior lower extremities (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 4 | 5
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal bloating (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 1 | 3 | 3
Diarrhea (Gastrointestinal disorders) | 5 | 1 | 5 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 2 | 0 | 1
Mucositis/stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Steatorrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 2 | 5 | 4
Oral pain (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 1 | 4 | 2
Jaundice (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal swelling after eating (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Peristalsis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ventral herniaexact (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 3 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Thrush (Candidiasis) (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Right sided bicep tear (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alkaline phosphatase (Investigations) | 4 | 3 | 2 | 5
ALT, SGPT (serum glutamic pyruvic transaminase) atinine (Investigations) | 6 | 4 | 6 | 7
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 5 | 4 | 3 | 10
Bilirubin (hyperbilirubinemia) (Investigations) | 4 | 2 | 0 | 0
Cholesterol high (Investigations) | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 2 | 3
GGT increased (Investigations) | 1 | 1 | 0 | 0
INR increased (Investigations) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 5 | 2 | 4 | 7
Lymphocyte count increased (Investigations) | 0 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 5 | 2 | 3 | 5
Platelet count decreased (Investigations) | 5 | 2 | 3 | 6
Weight loss (Investigations) | 1 | 2 | 0 | 3
White blood cell decreased (Investigations) | 6 | 2 | 4 | 4
Pneumatosis (Investigations) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 0 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 | 3 | 1 | 2
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 | 0 | 2 | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 | 1 | 2 | 2
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 | 5 | 5 | 10
Glucose, serum-low(hypoglycemia) (Metabolism and nutrition disorders) | 0 | 1 | 1 | 3
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Magnesium, serum-low(hypomagnesemia) (Metabolism and nutrition disorders) | 1 | 2 | 1 | 3
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 | 1 | 4 | 3
Potassium, serum-high(hyperkalemia) (Metabolism and nutrition disorders) | 1 | 0 | 2 | 5
Potassium, serum-low(hypokalemia) (Metabolism and nutrition disorders) | 2 | 4 | 0 | 2
Sodium, serum-high(hypernatremia) (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Sodium, serum-low(hyponatremia) (Metabolism and nutrition disorders) | 5 | 4 | 3 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Proteincalorie malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Low BUN (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Low chloride (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
High chloride (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Low serum protein (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Right maxilla met biopsied (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 5 | 0 | 2 | 2
Dysgeusia (Nervous system disorders) | 2 | 1 | 4 | 1
Headache (Nervous system disorders) | 6 | 1 | 2 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Anisocoria (Nervous system disorders) | 1 | 0 | 0 | 0
Attention deficit disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 2 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 2 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Intermittent mild cramping hands/feet (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Leg cramps at night (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 1 | 0 | 2 | 0
Flashing lights (Eye disorders) | 1 | 0 | 0 | 0
Scleral disorder (Eye disorders) | 1 | 0 | 0 | 0
Floaters (Eye disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Visual changes (Eye disorders) | 0 | 0 | 1 | 0
Decreased visual Acuity (Eye disorders) | 0 | 0 | 1 | 0
Urinary burning (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 1 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urine frequency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hot flashes (Vascular disorders) | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 2 | 1 | 1
Flushing (Vascular disorders) | 1 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
On review of the phase II data it was determined that the study did not meet continuation criteria according to Simon II stage design and would not meet criteria even with the remaining slot filled. The study was closed to further accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT01465659/Prot_SAP_000.pdf